CLINICAL TRIAL: NCT02025413
Title: Isolation of Circulating Tumor Cells Using a Novel EMT-Based Capture Method
Acronym: CTC-EMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Prostate Cancer Foundation (Other); United States Department of Defense (U.S. Federal Agency); Janssen Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Pro00032772
Record Dates: First submitted 2013-12-19; First posted 2014-01-01 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Metastatic Progressive Castration-resistant Prostate Cancer; Metastatic Progressive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metastatic progressive castration-resistant prostate cancer (Other): Mesenchymal-marker based ferrofluid (N-cadherin or O-cadherin based)
  Interventions: Device: Mesenchymal-marker based ferrofluid (N-cadherin or O-cadherin based)
- Metastatic progressive breast cancer (Other): Mesenchymal-marker based ferrofluid (N-cadherin or O-cadherin based)
  Interventions: Device: Mesenchymal-marker based ferrofluid (N-cadherin or O-cadherin based)

INTERVENTIONS:
Device: Mesenchymal-marker based ferrofluid (N-cadherin or O-cadherin based)

SUMMARY:
The primary objective of the preliminary lead-in study is to determine whether circulating tumor cells in patients with metastatic progressive castration-resistant prostate cancer or metastatic progressive breast cancer can be captured using a novel mesenchymal-marker based ferrofluid (N-cadherin or O-cadherin based).

The primary objective of each comparative cohort (second stage, prostate cancer) is to compare the non-detection rate of circulating tumor cells between the standard and novel methods.

ELIGIBILITY:
Inclusion Criteria:

Prostate cancer patients will be eligible for inclusion in this study only if all of the following criteria apply:

1. Histologically confirmed diagnosis of adenocarcinoma of the prostate. Small cell or neuroendocrine tumors of the prostate are also permitted.
2. Clinical or radiographic evidence of metastatic disease.
3. Castrate levels of testosterone (<50 ng/dl)
4. Evidence of disease progression on or following most recent therapy as evidenced clinically by the treating physician or by either of the following:

   * Two consecutive PSA levels greater than the PSA nadir achieved on ADT, separated by greater than one week
   * Radiographic evidence of disease progression as defined by new bone scan lesions or growth of soft tissue/visceral metastases >1 cm in diameter (2 cm for lymph nodes).
5. Age > 18 years.
6. Ability to understand and the willingness to sign a written informed consent document.

Breast cancer patients will be eligible for inclusion in this study only if all of the following inclusion criteria apply:

1. Histologically confirmed diagnosis of invasive breast cancer.
2. Clinical or radiographic evidence of metastatic disease.
3. Evidence of disease progression on the current or following the most recent therapy, determined either clinically by the treating physician or by radiographic evidence as defined by new bone scan lesions or soft tissue/visceral metastases >1 cm in diameter (2 cm for lymph nodes).
4. Age > 18 years.
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

1. History of intercurrent or past medical or psychiatric illness that would make participation in a blood drawing protocol difficult or not feasible at the discretion of the principal investigator or co-investigator(s).
2. Treatment with an anthracycline or mitoxantrone within 1 week of CTC collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by successfully detecting at least one CTC in at least 2 out of 10 subjects, comparing the non-detection rate over time. | The change in non-detection rate will be measured by comparing samples from Screening, Cycle 3, and Progression (up to 3 years)

SECONDARY OUTCOMES:
Comparison of the proportion of patients with no detectable CTCs between capture methods over time | Change will be measured by comparing samples at Screening, Cycle 3, Progression (up to 3 years)
Changes in CTCs (using each method) over time during systemic therapy | Screening, Cycle 3, Progression (up to 3 years)
Change in correlation of CTC enumeration using each method with baseline clinical and pathologic disease characteristics (for example, clinical stage, site of metastatic disease, Gleason sum for CRPC, PSA for CRPC, previous therapies) | Screening, Cycle 3, Progression (up to 3 years)
Median number of CTCs detected by each method over time | Changes will be measured from screening, cycle 3 and progression (up to 3 years)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Armstrong, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States